CLINICAL TRIAL: NCT06057532
Title: Impact of Carbohydrate Ingestion Prior to Urologic Surgery to Improve Patient Outcomes
Brief Title: Carbohydrate Ingestion Prior to Surgery (CIPS)
Acronym: CIPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jill Hamilton-Reeves, PhD RD LD, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00150605
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Urologic Surgical Procedures; Carbohydrate Loading; Preoperative Care
Keywords: Urologic Surgery; Preoperative Care; Carbohydrate Loading; Continuous glucose monitor
MeSH Terms: interventions — gatorade

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double-blinded, clinical trial that will provide a starch or standard sports drink at least 2 hours before surgery to evaluate perioperative glycemic variability. Patients will be randomized and have a 50/50 chance of getting one of the two drinks being studied.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drink powders will be measured and assigned a code by study staff that will not dispense the study drink powders to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UCAN SuperStarch study drinks (Experimental): Intervention group will receive UCAN SuperStarch study drinks. 100g carbohydrate will be consumed the night before surgery and 50g carbohydrate will be consumed 2 - 3 hours before surgery.
  Interventions: Dietary Supplement: UCAN SuperStarch
- Gatorade study drinks (Active Comparator): Active Control group will receive Gatorade study drinks. 100g carbohydrate will be consumed the night before surgery and 50g carbohydrate will be consumed 2 - 3 hours before surgery.
  Interventions: Dietary Supplement: Gatorade

INTERVENTIONS:
Dietary Supplement: UCAN SuperStarch — Intervention patients will have a continuous glucose monitor placed on their upper arm by the study team 1 - 5 days prior to surgery. These patients will drink the intervention study drink and record information about how they feel before and after consumption.
  Arms: UCAN SuperStarch study drinks
Dietary Supplement: Gatorade — Active control patients will have a continuous glucose monitor placed on their upper arm by the study team 1 - 5 days prior to surgery. These patients will drink the active control study drink and record information about how they feel before and after consumption.
  Arms: Gatorade study drinks

SUMMARY:
The objective is to determine the impact of taking a specialized form of carbohydrate in the immediate preoperative period on metabolic markers, surgical outcomes and patient health. Patients will be randomized to receive a specialized sports drink or a standard sports drink. Patients will have a continuous glucose monitor (CGM) placed on their upper arm to measure glucose throughout surgery and during the post-operative period.

DETAILED DESCRIPTION:
About 50 million major surgeries are performed annually in the United States. Longer duration surgeries increase metabolic demand and impose a greater risk of infections and worse outcomes than shorter duration surgeries. The release of hormones and catecholamines from surgery dampens the body's response to insulin which leads to acute insulin resistance. Even though the insulin resistance eventually resolves within weeks of surgery, metabolic stress during that window of time makes patients susceptible to infection and tissue catabolism. Therefore, there is a critical need to improve perioperative management of high-risk patients to decrease complications associated with major surgery which remains a significant cause of morbidity and mortality in these patients.

Up to 40% of patients undergoing major operations experience perioperative hyperglycemia (>140 mg/dL). Perioperative hyperglycemia has been implicated in increasing risk of perioperative complications including surgical site infection, reoperation, and mortality. With 50 million surgeries performed each year, preoperative optimization is essential for favorable postsurgical outcomes. A long-held dogma of prolonged fasting prior to the administration of anesthesia has slowed the adoption of consumption of carbohydrate drinks before surgery despite data showing a lower surgical stress response and decreased insulin resistance along with improved patient satisfaction. Multidisciplinary consensus has been necessary to implement change. The Enhanced Recovery after Surgery (ERAS) Society has shifted practice to optimize multidisciplinary perioperative care and one main tenet includes preoperative carbohydrate loading. While the dose and type vary across institutions and practices, the American Society of Enhanced Recovery/Perioperative Quality Initiative joint consensus statement and the American Society of Anesthesiologists recommend consumption of a preoperative beverage containing ≥50 g of carbohydrate (CHO) for surgical patients 2-3 hours prior to surgery. Despite this recommendation, the practice of preoperative oral intake has still lagged with only 20% adherence in surgical care pathways.

ELIGIBILITY:
Inclusion Criteria:

* adults, at least 18 years old,
* undergoing major urologic surgery (proposed duration more than 4 hours),
* must be able to swallow liquid,
* must speak English.

Exclusion Criteria:

* diagnosis of Type 1 or 2 diabetes mellitus
* A1C of 6.5% or higher
* pregnant or lactating
* known allergy to milk, soy, egg, wheat, peanuts, tree nut,
* swallowing difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Compare perioperative glycemic variability between study arms | From up to 5 days before surgery to up to 4 days after surgery.
  Differences in blood glucose, insulin, free fatty acids will be compared
Compare perioperative clinical outcomes after surgery between study arms | From surgery to 90 days after surgery.
  Differences in post-operative complications within 30 days after surgery, length of hospital stay, post-operative infections, and number of patients needing intraoperative or postoperative insulin treatment will be be compared between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Hamilton-Reeves, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Health System, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dobson GP. Trauma of major surgery: A global problem that is not going away. Int J Surg. 2020 Sep;81:47-54. doi: 10.1016/j.ijsu.2020.07.017. Epub 2020 Jul 29. PMID 32738546
- [Background] Cheng H, Clymer JW, Po-Han Chen B, Sadeghirad B, Ferko NC, Cameron CG, Hinoul P. Prolonged operative duration is associated with complications: a systematic review and meta-analysis. J Surg Res. 2018 Sep;229:134-144. doi: 10.1016/j.jss.2018.03.022. Epub 2018 Apr 24. PMID 29936980
- [Background] Thorell A, Loftenius A, Andersson B, Ljungqvist O. Postoperative insulin resistance and circulating concentrations of stress hormones and cytokines. Clin Nutr. 1996 Apr;15(2):75-9. doi: 10.1016/s0261-5614(96)80023-9. PMID 16844002
- [Background] Kielhorn BA, Senagore AJ, Asgeirsson T. The benefits of a low dose complex carbohydrate/citrulline electrolyte solution for preoperative carbohydrate loading: Focus on glycemic variability. Am J Surg. 2018 Mar;215(3):373-376. doi: 10.1016/j.amjsurg.2017.10.029. Epub 2017 Nov 8. PMID 29128103
- [Background] Ackerman RS, Tufts CW, DePinto DG, Chen J, Altshuler JR, Serdiuk A, Cohen JB, Patel SY. How Sweet Is This? A Review and Evaluation of Preoperative Carbohydrate Loading in the Enhanced Recovery After Surgery Model. Nutr Clin Pract. 2020 Apr;35(2):246-253. doi: 10.1002/ncp.10427. Epub 2019 Oct 21. PMID 31637778
- [Background] Nygren J, Soop M, Thorell A, Sree Nair K, Ljungqvist O. Preoperative oral carbohydrates and postoperative insulin resistance. Clin Nutr. 1999 Apr;18(2):117-20. doi: 10.1054/clnu.1998.0019. PMID 10459075
- [Background] Hausel J, Nygren J, Lagerkranser M, Hellstrom PM, Hammarqvist F, Almstrom C, Lindh A, Thorell A, Ljungqvist O. A carbohydrate-rich drink reduces preoperative discomfort in elective surgery patients. Anesth Analg. 2001 Nov;93(5):1344-50. doi: 10.1097/00000539-200111000-00063. PMID 11682427
- [Background] MENDELSON CL. The aspiration of stomach contents into the lungs during obstetric anesthesia. Am J Obstet Gynecol. 1946 Aug;52:191-205. doi: 10.1016/s0002-9378(16)39829-5. No abstract available. PMID 20993766
- [Background] Wischmeyer PE, Carli F, Evans DC, Guilbert S, Kozar R, Pryor A, Thiele RH, Everett S, Grocott M, Gan TJ, Shaw AD, Thacker JKM, Miller TE, Hedrick TL, McEvoy MD, Mythen MG, Bergamaschi R, Gupta R, Holubar SD, Senagore AJ, Abola RE, Bennett-Guerrero E, Kent ML, Feldman LS, Fiore JF Jr; Perioperative Quality Initiative (POQI) 2 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Nutrition Screening and Therapy Within a Surgical Enhanced Recovery Pathway. Anesth Analg. 2018 Jun;126(6):1883-1895. doi: 10.1213/ANE.0000000000002743. PMID 29369092
- [Background] Joshi GP, Abdelmalak BB, Weigel WA, Harbell MW, Kuo CI, Soriano SG, Stricker PA, Tipton T, Grant MD, Marbella AM, Agarkar M, Blanck JF, Domino KB. 2023 American Society of Anesthesiologists Practice Guidelines for Preoperative Fasting: Carbohydrate-containing Clear Liquids with or without Protein, Chewing Gum, and Pediatric Fasting Duration-A Modular Update of the 2017 American Society of Anesthesiologists Practice Guidelines for Preoperative Fasting. Anesthesiology. 2023 Feb 1;138(2):132-151. doi: 10.1097/ALN.0000000000004381. PMID 36629465
- [Background] Colebatch E, Lockwood C. Enhanced perioperative nutritional care for patients undergoing elective colorectal surgery at Calvary North Adelaide Hospital: a best practice implementation project. JBI Evid Synth. 2020 Jan;18(1):224-242. doi: 10.11124/JBISRIR-2017-003994. PMID 31290790